CLINICAL TRIAL: NCT06610461
Title: High-flow Nasal Oxygen Versus Face Mask or Nasal Cannula for Advanced Endoscopy in High-risk Patients
Brief Title: High-flow Nasal Oxygen Therapy for Advanced Endoscopy in High-risk Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Maximilian S Schaefer, Director of the Center for Anesthesia Research Excellence (CARE), Division Director of Thoracic Anesthesia, Assistant Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023P000245
Record Dates: First submitted 2024-08-30; First posted 2024-09-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Hypoxemia During Surgery
Keywords: Nasal cannula, humidified oxygen, hypoxemia, endoscopy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: This study will be a non-blinded, randomized, controlled trial comparing two study groups ("intervention" and "control"). Participants are assigned to one of two groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control group (No Intervention): Supplemental oxygen throughout anesthesia in accordance with hospital guidelines.
- Intervention group (Active Comparator): HFNO- treatment
  Interventions: Device: HFNO-Treatment

INTERVENTIONS:
Device: HFNO-Treatment — The investigated intervention is the application of HFNO throughout a high-risk upper GI-endoscopy. Concentration of oxygen is 100%. Prior to induction, flow rate is set to 20 l/min and increased to 30 l/min if tolerated by the patient. After induction of anesthesia, flow rate is increased to 60 l/min and maintained throughout the anesthesia.
  Arms: Intervention group

SUMMARY:
Anesthesia is crucial during upper GI endoscopy in order to improve the procedural conditions for the interventionist, increase the quality of examination and alleviate patient discomfort. However, sedation during endoscopy carries a serious risk of blood oxygen desaturation.

This study aims to investigate the hypothesis if the application of high-flow nasal oxygen (HFNO) during high-risk gastroscopy reduces the risk of blood oxygen levels to drop below a defined threshold. Enrolled patients will be randomly assigned to either the control group, receiving standard care during endoscopy, or the intervention group, receiving HFNO therapy during the procedure. Throughout the intervention, vital parameters will be recorded. Care providers will be asked to answer a questionnaire that specifically evaluates the effect of HFNO on patient safety and the procedure.

DETAILED DESCRIPTION:
This non-blinded, randomized controlled trial compares two study groups, the interventional and control group, to investigate whether HFNO-treatment reduces the risk of hypoxemia during peri-interventional high-risk upper GI endoscopy.

The randomization schema is developed by an unblinded statistician using SAS (Statistical system) and uploaded to the REDCap randomization module, enabling delegated team members to generate sequential allocations for enrolled subjects.

Patients assigned to the control group will receive supplemental oxygen throughout anesthesia in accordance with hospital guidelines, either using a standard nasal cannula or procedural oxygen mask (POM). The choice of supplemental oxygen delivery, as well as oxygen flow rates, are at the discretion of the anesthesia provider. Post-anesthesia, patients will be transferred to the recovery room with either the standard nasal cannula or procedural oxygen mask at a flow rate determined by the anesthesia provider.

Patients assigned to the intervention group will receive humidified oxygen throughout anesthesia in order to assess the effect of HFNO. High-flow nasal cannula (Fisher & Paykel Optiflow) are connected prior to induction of anesthesia, allowing for different flow rates and oxygen concentration to be administered according to the study protocol. The oxygen concentration of the delivered gas for the trial is 100%. Prior to induction, flow rate will be set to 20 liters per minute and increased to 30 liters per minute if tolerated by the patient. After induction of anesthesia, flow rate will be increased to 60 liters per minute and maintained throughout anesthesia. After anesthesia, the high-flow nasal cannula will be exchanged to a standard nasal cannula and the patient will be transferred to the recovery room at which point the flow rate will be determined by the anesthesia provider.

The decision to discontinue the intervention of the study is entirely at the discretion of the attending anesthesiologist. Alternative means of supplemental oxygen delivery, such as nasal cannula or oxygen mask, may be considered by the attending anesthesiologist. If the intervention is discontinued, the rationale for the decision is documented for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* Upper endoscopy (EGD, ERCP, EUC etc.) w/wo colonoscopy expected duration > 15 min under MAC

  * one or more of the following:
* Diagnosis of sleep apnea
* BMI ≥ 30 kg/m2
* Baseline SpO2 < 96% or Requirement for long-term oxygen therapy
* BOSTN score ≥ 2

  * BMI ≥ 30 kg/m2
  * Observed apnea
  * Observed loud Snoring
  * Daytime Tiredness
  * Neck circumference ≥ 16.5 inches in female, ≥ 17.5 inches in male

Exclusion Criteria:

* Known Pregnancy
* Known Current infection with COVID-19
* Planned general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Additional actions had to be taken to ensure sufficient SpO2 oxygenation. | The primary outcome will be assessed in the time between start of induction of anesthesia and awakening until discharge from the procedural room, which is typically between 30 and 120 minutes
  A composite outcome including the occurrence of any airway manipulation due to inadequate ventilation, which may include jaw thrust or Esmarch maneuver, bag-mask ventilation, insertion of a nasogastric tube, laryngeal mask airway or endotracheal intubation or procedural interruption to treat inadequate ventilation. The necessity for airway manipulation is at the discretion of the anesthesia provider. Documentation of the primary outcome is conducted on paper sheets by the anesthesia provider including time, type and reason of upper airway manipulation.

SECONDARY OUTCOMES:
Satisfaction of care provider | Satisfaction of the provider will be assessed at the end of the procedure upon discharge from the procedure room and will relate to the duration of the procedure, typically between 30 and 120 minutes
  Satisfaction of the endoscopist is assessed at the end of the procedure. Satisfaction is rated on a numeric rating scale from 0 to 10, zero being completely dissatisfied and 10 being completely satisfied.
Procedure interruption | Procedure interruption will be assessed for the duration of the procedure, which is typically between 30 and 120 minutes
  The occurrence of procedure interruption, defined as prompting the endoscopist to stop the procedure, or removal of the scope for treatment of inadequate ventilation.
Occurrence of hypoxemia | The occurence of hypexmia will be assessed in the time between start of induction of anesthesia and awakening until discharge from the procedural room, which is typically between 30 and 120 minutes
  It is determined as SpO2 <92% in the absence of obvious artefacts during anesthesia. Absence of artefacts is defined as the presence of a sinusoid plethysmography curve.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia, Critical Care and Pain Medicine Department at Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin OS. Sedation for routine gastrointestinal endoscopic procedures: a review on efficacy, safety, efficiency, cost and satisfaction. Intest Res. 2017 Oct;15(4):456-466. doi: 10.5217/ir.2017.15.4.456. Epub 2017 Oct 23. PMID 29142513
- [Result] Elphick DA, Donnelly MT, Smith KS, Riley SA. Factors associated with abdominal discomfort during colonoscopy: a prospective analysis. Eur J Gastroenterol Hepatol. 2009 Sep;21(9):1076-82. doi: 10.1097/MEG.0b013e32832357b3. PMID 19339891
- [Result] Ahrens E, Tartler TM, Suleiman A, Wachtendorf LJ, Ma H, Chen G, Kendale SM, Kienbaum P, Subramaniam B, Wagner S, Schaefer MS. Dose-dependent relationship between intra-procedural hypoxaemia or hypocapnia and postoperative delirium in older patients. Br J Anaesth. 2023 Feb;130(2):e298-e306. doi: 10.1016/j.bja.2022.08.032. Epub 2022 Oct 1. PMID 36192221
- [Result] Qadeer MA, Lopez AR, Dumot JA, Vargo JJ. Hypoxemia during moderate sedation for gastrointestinal endoscopy: causes and associations. Digestion. 2011;84(1):37-45. doi: 10.1159/000321621. Epub 2011 Feb 8. PMID 21304242
- [Result] Lenglet H, Sztrymf B, Leroy C, Brun P, Dreyfuss D, Ricard JD. Humidified high flow nasal oxygen during respiratory failure in the emergency department: feasibility and efficacy. Respir Care. 2012 Nov;57(11):1873-8. doi: 10.4187/respcare.01575. Epub 2012 Mar 13. PMID 22417844
- [Result] Nay MA, Fromont L, Eugene A, Marcueyz JL, Mfam WS, Baert O, Remerand F, Ravry C, Auvet A, Boulain T. High-flow nasal oxygenation or standard oxygenation for gastrointestinal endoscopy with sedation in patients at risk of hypoxaemia: a multicentre randomised controlled trial (ODEPHI trial). Br J Anaesth. 2021 Jul;127(1):133-142. doi: 10.1016/j.bja.2021.03.020. Epub 2021 Apr 28. PMID 33933271
- [Result] Mazzeffi MA, Petrick KM, Magder L, Greenwald BD, Darwin P, Goldberg EM, Bigeleisen P, Chow JH, Anders M, Boyd CM, Kaplowitz JS, Sun K, Terrin M, Rock P. High-Flow Nasal Cannula Oxygen in Patients Having Anesthesia for Advanced Esophagogastroduodenoscopy: HIFLOW-ENDO, a Randomized Clinical Trial. Anesth Analg. 2021 Mar 1;132(3):743-751. doi: 10.1213/ANE.0000000000004837. PMID 32398433